CLINICAL TRIAL: NCT05015777
Title: Effects of Jaques-Dalcroze Eurhythmics Program on Postural Stability in Elderly Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1/16
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Aging Problems; Coordination Impairment
Keywords: postural stability; elderly; Dalcroze Eurhythmics; center of pressure; biofeedback
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Intervention Model Description: A study model based on randomized controlled trial - parallel group design was used.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Those conducting the measurements were unaware of the purpose of this study and the fact that the participants were divided into groups

ARMS (2):
- Intervention Group (Experimental): Participated in the exercise programme
  Interventions: Other: Emil Jaques-Dalcroze's Eurhythimcs Exercise Program
- Control Group (No Intervention): Were advised not to change anything about their current lifestyle, and in particular not to undertake any new structured physical activity.

INTERVENTIONS:
Other: Emil Jaques-Dalcroze's Eurhythimcs Exercise Program — Training sessions took place twice a week for 45 minutes each over a period of 12 weeks. Each training included rhythmic exercises using the Jaques-Dalcroze Eurhythmics (JDE) method with piano accompaniment and electronically played music. Training sessions were conducted by a JDE specialist.
  Exercises with the use of this method consist mainly in the repetition of preset musical sequences using body movements. In addition to the physical layer, the cognitive layer was equally important: while performing a given movement exercise, participants often had to focus in order to react appropriately to additional tasks, such as changes in sound pitch and rhythm of the piece.
  Arms: Intervention Group

SUMMARY:
This study investigated the effect of exercise using the Emil Jaques-Dalcroze's method on the postural stability of women over 65 years of age. The study model was based on a randomized controlled trial - parallel group design.

DETAILED DESCRIPTION:
Participants were recruited through advertisements in local newspapers and on the Internet, and covered the Poznań Metropolitan Area, Poland. Following randomization using the computer program Statistica 13.4 (TIBCO Software Inc., Palo Alto, CA)., the participants were divided into two groups: Intervention Group (IG) and Control Group (CG). The participants' postural stability was investigated by determining their ability to control the displacement of the body's center of pressure (COP). For this purpose, the Balance Platform model AccuSway Plus was used, together with the Balance Trainer software. The system recorded changes in COP position in the anteroposterior (AP) and mediolateral (ML) directions. The sampling rate was set at 100 Hz. The COP is a reliable parameter for evaluating postural stability and upright balance control. The results of the four COP parameters described below were statistically analysed.

1. COP Path Length: sum of path lengths from the Subject Start Position to the intersection of the active target perimeter.
2. COP Area Deviation: sum of areas where the COP path deviates from the straight line that intersects the Subject Start and End Positions.
3. COP Total Time: time taken to complete the entire trial.
4. COP Reaction Time: average reaction time to cross the perimeter of target, measured from the activation of the next target.

Two measurement sessions were held: the first (baseline) took place during the week before starting the exercise programme and the second (12-week follow-up) straight after its finish. Women with IG participated in the exercise programme, while women with CG were advised not to change anything about their current lifestyle, and in particular not to undertake any new structured physical activity. Those conducting the measurements were unaware of the purpose of this study and the fact that the participants were divided into groups.

Training programme. Training sessions took place twice a week for 45 minutes each over a period of 12 weeks. Each training included rhythmic exercises using the Jaques-Dalcroze Eurhythmics (JDE) method with piano accompaniment and electronically played music. Training sessions were conducted by a JDE specialist.

Balance Platform Test Participants had to perform a movement task while standing on a posturographic platform. A Feedback Balance Analysis protocol was used - the subjects saw a point on the screen that was a reflection of their COP. By tilting their body in different directions, they could observe changes in the position of their COP in real time. The participants' task was to do it in such a way as to direct their COP to the appropriate targets marked on the screen, in the right order.

Taking into account the natural heterogeneity of the group in terms of physical fitness due to the age of subjects, the distances of extreme areas in relation to the central area, and thus the range of deflection, were decided to be determined for each participant individually. For this purpose, first the maximum deflections of each subject in the AP and ML directions were determined, and then the software automatically determined the centres of targets at a distance of 75% of the maximum deflection in a given direction. This ensured that each subject leaned their torso relatively the same range and that the task was within their capabilities. The results of maximum torso lean ranges were also statistically analysed.

The test consisted of two main elements: 1) the COP point movement phase and 2) the COP point maintain phase. The task consisted of the COP point movement to individual targets (in a predetermined order), each time the COP point had to be maintained inside the area of each target for at least one second, after which the target became inactive (darker), which was a signal of its correct passing. At the same time, the next (active) target would light up, indicating that the COP point had to be moved to that target, where it again had to be held for a minimum of one second, and so on. Each time the extreme target was passed, it was necessary to return to the central target. A similar trial measuring changes in postural stability in a biofeedback model under the influence of training has already been used in other experiments.

The posturographic platform was fixed to a flat surface, in front of the subject at a distance of 1.5 meters at eye level was placed a 27 inch monitor. The room was soundproofed to ensure peace and quiet. On the platform there were lines specifying the proper distances and angles of feet placement in order to ensure that the subject stood in the same place during each subsequent trial. The feet on the platform were placed naturally, one next to the other at hip width, with the toes gently pointing outwards.

Each participant was given verbal instructions on how to perform the test, with particular emphasis on the fact that the test had to be carried out as quickly and accurately as possible, moving the COP point by the shortest possible route to the target, and once reached, trying to keep the COP point as still as possible in the centre of target until it became inactive (turned dark). The person conducting the test next performed a demonstration of the entire trial. The final step was for the subjects to perform two pre-test trials, followed by a third trial, the results of which were statistically analysed.

Statistical analysis The results of descriptive statistics were presented as means with standard deviation (mean±SD). Postural stability test results were presented as means and confidence intervals at the 95% level. A two-factor analysis of variance (ANOVA) was conducted. An eta square analysis was used to determine effect size. The post-hoc Tukey test was conducted in case of significant main or interaction effects. Differences between groups in the single study session area and between study sessions in the group area were determined using the Mann-Whitney U test with correction for continuity. Statistical significance level was set at 5%. All calculations were carried out using Statistica 13.4 (TIBCO Software Inc., Palo Alto, CA).

ELIGIBILITY:
Inclusion Criteria:

* women,
* community-dwelling,
* had no contraindications to participation in physical activity,
* scored at least 8 on the Abbreviated Mental Ability Test .

Exclusion Criteria:

* taking medications that may interfere with natural control of postural stability,
* users of orthopaedic equipment,
* patients with neurological disease (Parkinson's or Alzheimer's),
* patients with significant visual and/or auditory perception impairment,
* subjects who undertake or have undertaken regular physical activity in the past three years

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-03-06 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Ability to control the displacement of the body's center of pressure (COP). | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JAN ADAMCZYK, MA, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan, Poland